CLINICAL TRIAL: NCT05784116
Title: Immune/Inflammatory Biomarkers in Postpartum Depression: Pathogenetic Mechanisms, MRI Endophenotypes, and Predictive Biomarkers
Brief Title: Immune/Inflammatory Biomarkers in Postpartum Depression
Acronym: PPDINFLAME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Francesco Benedetti, Group Leader, IRCCS San Raffaele
Other Study IDs: RF-2019-12371066
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum, Peripheral whole blood for gene expression, PBMC cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This will be a very straightforward study assessing changes of immune/inflammatory peripheral biomarkers before/after delivery with postpartum mood and the psychopathological features of postpartum depression (PPD), and with MRI measures of functional and structural brain integrity.

Multimodal assessment of peripheral cytokines, PBMC gene expression, FACS immunophenotyping, and IDO activation, will be validated with (a) clinical data about the presentation of PPD, (b) self- and observer ratings of psychopatology, (c) results coming from neuropsychological assessment of cognitive functions, and (d) multimodal brain imaging outcomes (WM integrity, functional connectivity, GM volumes).

It is expected that worsening or stabilization of mood, and the diagnosis of PPD, will be paralleled by worsening or stabilization of these measures, thus providing new markers to estimate the susceptibility to the disorder, to identify targets for treatment, and to predict and monitor treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

-Signed informed consent, able to understand, speak and write the national language

Exclusion Criteria:

* History of bipolar disorder, schizophrenia, schizoaffective disorder, psychosis NOS; anorexia or bulimia nervosa;
* Taking following medications: antipsychotics, anticonvulsants, mood stabilizers, stimulants
* Active infection requiring antibiotics therapy;
* Immunosuppressed patient
* Other chronic diseases
* Signs of active infection requiring treatment
* Use of anti-inflammatory medication on a regular basis for a chronic inflammatory/autoimmune Disorder. - - Forbidden treatment: corticosteroids, NSAD, immunosuppressant IV-Ig based treatment
* Ongoing fever, infection treated by antibiotics or uncontrolled diabetes type I or II;
* Existing cancer or history of cancer in the last 5 years (except skin epidermoid cancer or in-situ cervix cancer);
* Known HIV infection or clinically manifest Acquired Immune Deficiency Syndrome (AIDS), Parkinson's or Alzheimer's disease, or any other serious condition likely to interfere e with the conduct of the trial;
* Abuse of drugs or alcohol in the past 6 months
* Presence of chromosomal disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 150 pregnant women will be recruited in each center. We expect 15-30 women per group to develop PPD and be matched with HC in a 1:2 ratio, yielding a sample of 30-60 PPD patients and 60-120 HC.
  Patients will be recruited at the Department of Obstetrics and Ginecology of Ospedale San Raffaele and at the Department of Woman, Children and Newborn (Clinica Mangiagalli), Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico.
  Patients will be recruited at the 20th week of gestation when patients fulfilling the inclusion criteria will be offered the possibility to participate to the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-11-24 (Estimated); Study Completion 2024-11-24 (Estimated)

PRIMARY OUTCOMES:
Peripheral inflammation | 9 months
  peripheral markers of immune/inflammatory activation before/after delivery predicting pre- and post-partum depressive psychopathology
Postpartum depression | 9 months
  condition of PPD in the six months following delivery

SECONDARY OUTCOMES:
Multimodal MRI | 9 months
  To correlate peripheral markers of immune/inflammatory activation with multimodal MRI measures of WM and GM integrity, functional connectivity, 1H-MRS spectroscopy, and with measures of cognitive functions in PPD

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Benedetti, MD, Principal Investigator — IRCCS Ospedale San Raffaele, Milano
Locations (1):
- Ospedale San Raffaele, Milan, Italy